CLINICAL TRIAL: NCT04258852
Title: Understanding Factors That Influence Electronic Cigarette Nicotine Delivery Through PET Imaging of Beta-2 Nicotinic Acetylcholine Receptors
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment halted by pandemic
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2000023604; 1K23DA045957-01 (NIH)
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Electronic Cigarette Use
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Strength, High Strength (Experimental)
  Interventions: Drug: Low strength nicotine e-liquid; Drug: High strength nicotine e-liquid
- High Strength, Low Strength (Experimental)
  Interventions: Drug: Low strength nicotine e-liquid; Drug: High strength nicotine e-liquid

INTERVENTIONS:
Drug: Low strength nicotine e-liquid — Low strength nicotine e-liquid
Drug: High strength nicotine e-liquid — High strength nicotine e-liquid

SUMMARY:
The goal of this proposal is to test the overall hypothesis that e-cigarettes (ECs) provide efficient nicotine delivery to the brain and arterial blood in non-EC-naïve smokers and e-cigarette users and that EC liquid characteristics modulate this effect. This study will test the hypothesis through complementary methods that include [ [18F]NCFHEB (aka [18F]Flubatine) PET neuroimaging, arterial blood nicotine measurements, and subjective drug effects assessments.

DETAILED DESCRIPTION:
C.2 Subject Inclusion and Assessments Overall study design: Non-EC-naïve smokers or e-cigarette users (n=20) will abstain from tobacco smoking/nicotine products for 5 days prior to each PET scan. In a randomized order (counterbalanced), after baseline quantification of receptor availability, subjects will be scanned while using an EC: (1) "JUUL" 5%, a common commercially available unmodified nicotine salt EC, and (2) JUUL 3%, a lower nicotine strength product. A third optional scan where subjects smoke a cigarette may be conducted but is not required. During scanning, subjects will undergo arterial blood nicotine level measurements following EC use and measures of nicotine withdrawal, craving, and drug effects will be measured. 5-7 days of smoking abstinence will be required prior to each PET scan to ensure no residual nicotine occupies receptors. Subjects will go back to smoking as usual after first scan for 2-3 weeks prior to subsequent smoking abstinence/PET scanning. Subjects will be provided with smoking cessation resources upon request.

C.2.b Subjects: Twenty non-EC-naïve tobacco dependent smokers or e-cigarette users will be recruited for the study. All research subjects will be recruited under guidelines of the Yale University Institutional Review Board (Human Investigation Committee). Smokers will be recruited from the community via IRB-approved advertising. After completing informed consent, subjects will have a psychiatric, physical and neurological examination, laboratory tests and an electrocardiogram (EKG) (see C.2.c Clinical Assessments below). This is considered the screening phase. Subjects will be excluded for major medical, neurological or psychiatric illness, abnormal laboratory tests, or contraindication to PET or MR imaging. A urine drug screen and pregnancy test are performed at screening and prior to each imaging session and participants are excluded for a positive test. Detailed inclusion/exclusion criteria can be found in Protection of Human Subjects section. All women will be required to have a negative urine pregnancy test and all subjects are required to have a negative urine drug toxicology test prior to radiotracer administration.

C.2.c Clinical Assessments: A standardized battery will be administered to all subjects at intake including Health Questionnaire, the SCID, assessments of demographics, measures of tobacco use, alcohol and drug use, family history of smoking, mood (PROMIS short forms for depression, anxiety, and anger), Center for Epidemiologic Studies Depression Scale), anxiety (State Trait Anxiety Inventory), impulsivity (Brief - Barratt Impulsivity Scale, smoking dependence (PROMIS nicotine dependence scale), smoking craving (Tiffany QSU) and withdrawal (Minnesota Nicotine Withdrawal Scale). Mood and smoking assessments will be repeated on each scan day before and after challenge. Product liking, craving and the Drug Effects Questionnaire (DEQ) will be assessed on a subjective scale (0-100, low-high) immediately following product use. The DEQ will measure acute effects consisting of seven items: drug strength, high, feeling stimulated, good effects, bad effects, wanting more drugs, and drug liking.

Baseline and after each PET scan/e-cig challenge:

* Health Questionnaire
* PROMIS Dyspnea Severity Item Pool
* PROMIS Dyspnea Characteristics
* PROMIS Fatigue Short Form
* Functional Assessment of Chronic Illness Therapy (FACIT) Cough item
* The health questionnaire titled 'assessment of health problems' (and provided as an attachment via a comment in IRES) will be added to the protocol and will be completed at intake and before each exposure. Note that potential subjects with chronic symptoms that would interfere with monitoring of vaping complications, will not be enrolled.

Positive findings of a change in symptom or single severe symptom would trigger clinical referral to a treating physician or the emergency room.

C.2.d Contingency Management: All smokers/e-cigarette users will be helped to remain abstinent for 5- 7 days prior to each PET scan with highly successful contingency management techniques that have been used extensively in the laboratory before. Subjects will return to smoking use as usual after the first PET scan and repeat smoking abstinence prior to the next PET scan. This technique has been successful in the past to study nicotine occupancy of receptors after multiple challenges by recruiting smokers who are non-treatment seeking. Subjects will be met daily over the course of abstinence provide support and obtain CO and urine cotinine levels to ensure smoking abstinence. Subjects who are not able to abstain from tobacco smoking (2 consecutive days without a decrease in urine cotinine levels or a sudden increase in urine cotinine or CO levels) will be withdrawn from the study.

C.2.e - MRI/cognitive testing Subjects will be asked to go to the MRRC at The Anlyan Center for Medical Research & Education (TAC, 300 Cedar Street) to have an MRI (Magnetic Resonance Imaging) scan of their brain. The purpose of the MRI is to help us identify the different regions of their brain on the PET scans.

The MRI scan is a routine way to get pictures of the inside of the body. Subjects will be asked if they are carrying any metallic objects before they move toward the MRI system. These objects will be held for them in a locked cabinet in the MRI Center to avoid having these objects fly toward the magnet when they approach it. They will also be asked to walk through a metal detector. They will be asked to lie still in the MRI scanner for about 30 minutes. The scanner looks like a deep tunnel. They will be inside the tunnel from head to knees. They will not be able to see out of it, but they will be able to hear us and be heard if they wish to say anything. They will hear a drumming noise when the camera is taking pictures of their brain. If they feel uncomfortable during the scan, the scan will be ended at any time they wish. However, if they cannot complete the MRI scan, they will not be able to participate in any more of these studies.

Two sessions of testing of their memory, attention, and concentration may take place. This will take approximately 1hr total. They will be given a break between these sessions. This may take place on the same day as the MRI scan, or on another day prior to PET scans if that works better with their and staff schedule.

During this visit, they may play a computer game called the Face Game. The goal of the Face Game is to win as much money as possible. They may earn money by quickly and correctly pressing one of two keys on the keyboard, each time they see a face on the screen. They will press one key if they think that the mouth on the face is long, and the other if they think it is short.

Cold Pressor Task Subjects may also be asked to participate in the cold pressor task during the study to test the body's physiological response to cold water. They will be asked to immerse your hand in a bucket of ice cold water maintained at 0-4°C. They will be told to raise their other hand when they begin to feel pain and to remove their hand from the water when they can no longer tolerate the pain. While their hand is immersed in water, they will also be asked to rate their pain on a scale from 0-100 and their heart rate and blood pressure will be monitored.

Impulsivity Subjects may be asked to play a game in which they will use a computer mouse to click a balloon pump that inflates a balloon on the screen. The objective of the task is to get the largest amount of the money possible while avoiding balloon explosions. This assessment tests their impulsivity. They may be asked to play this game on the day of their PET scan too.

C.3. PET Imaging Procedures PET procedures will be conducted at the Yale University PET Center. Female subjects will be given a urine pregnancy test prior to the initiation of any imaging procedures. If the test is positive, the scans will be canceled. Subjects will receive a minimum of 2 and maximum of 3 PET scans. The 3rd scan is optional.

PET scans: Prior to the PET scans, a T1-weighted MRI will be acquired for all subjects on a 3.0 Tesla Siemens Trio camera to rule out any brain abnormalities and for anatomical reference in the image analysis.

PET scans are acquired as subjects lie supine on the scanner bed. Venous catheters will be used for intravenous administration of the radiotracer, and possibly for additional venous blood sampling. A radial artery catheter will be inserted by an experienced physician before the PET scan to draw arterial blood samples for metabolite analysis and for determination of the fraction of plasma radioactivity unbound to protein.

Infusion of the radiotracer takes 210 minutes (3.5 hours). Subjects will be scanned for 2 hours (starting 90 minutes after initiation of radiotracer infusion).

[18F]NCFHEB will be synthesized and administered on PET scan days as a bolus plus constant infusion with a Kbol of 360 minutes over 3.5 hours. PET data will be acquired on the MCT. A 6-min transmission scan will be acquired at the beginning or end of each PET scan to correct for attenuation. Arterial blood samples will be taken to obtain a metabolite-corrected [18F]NCFHEB input function. Baseline receptor availability will be measured 90-120mins after radiotracer infusion. Then, subjects will start a challenge (NIDA EC or JUUL EC, counterbalanced order) at 125min for 5 minutes in the scanner. Thereafter, post nicotine scanning will continue until end of 4 hrs of infusion. Vital signs (blood pressure, pulse, respiration) and ECG's will be obtained before and after radiotracer administration. The same procedures will follow for the 2nd PET scan.

Use of EC: Subjects will receive 2 different scans and will puff one of two EC products (in random order, counterbalanced): "JUUL" 5% (50 mg/ml), a common commercially available unmodified nicotine salt EC, and (2) JUUL 3% (30 mg/ml), a lower nicotine strength product. Only tobacco flavor will be used. A training session to familiarize smokers with the EC product used in the study will be conducted at an appointment prior to the PET scans. Subjects will be advised to take longer and slower puffs from the EC (at least 3-4 seconds) as compared with puffing a cigarette. During each scan, subjects will be instructed to puff on the EC for up to 5 minutes. All users will be directly observed during EC use to ensure they do not have any problems operating the device. If available, a mouthpiece to measure puff topography may be used as previously described.

Use of Regular Cigarette: A third PET scan using a regular cigarette may be offered for cigarette smokers but is not required for study completion.

Blood Samples: On PET scan days, arterial blood samples will be collected prior to radiotracer administration and at multiple time points (t = 0, 0.3, 1, 3, 5, 10, 20, 30, 60, 90 minutes post challenge) after EC/cigarette use to determine nicotine concentrations in the blood, which will be assayed using liquid chromatography tandem-mass spectrometry with deuterated internal standards.47 These data will be used to calculate pharmacokinetic patterns of nicotine delivery under each condition (Cmax, Tmax, and AUC for nicotine).

Image Analysis and Outcome Measure: List-mode PET data will be reconstructed with OSEM with built-in corrections for attenuation, normalization, scatter, randoms, deadtime and subject motion.53,54 Following image reconstruction, a summed image will be registered to the subject's MRI. Regions of interest (ROIs) will be anatomically defined using a template [Anatomical Automatic Labeling (AAL)] coregistered to the subject's MRI image. ROIs used for calculation of receptor occupancy will be: cerebellum, frontal, parietal, temporal, and occipital cortices, caudate, putamen, hippocampus, and amygdala. These regions are chosen because they were previously examined in β2*-nAChR studies, have significant density in the human brain, and are relevant to the craving and withdrawal properties of nicotine. The thalamus will not be included because equilibrium is not reached in this region with the bolus-infusion paradigm. The volume of distribution VT will be estimated using the equilibrium ratio between total radioactivity concentration in tissue and parent concentration in arterial plasma. Baseline VT will be estimated from 90-120 min after infusion start, previously shown to establish good equilibrium in brain Post-ECig VT will be estimated from 180-210 minutes after infusion start (55-85 minutes post challenge). Prior preliminary data show that this is a sufficient amount of time for a new steady state to be achieved. Receptor occupancy and VND will be estimated using the Lassen plot approach.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, aged 21-55 years
* Able to read and write English
* Able to give voluntary, written informed consent
* Current cigarette smoking or e-cigarette use
* Non-treatment seeking
* Exhaled CO > 10 ppm or urine cotinine > 50 ng/ml
* Agreement to only use e-cigarette products provided in the study
* Not naïve to vaping (3 or more months and 12 or more times).

Exclusion Criteria:

* Current medical condition such as neurological, pulmonary, cardiovascular, endocrine, renal, liver, or thyroid pathology
* History of or current neurological or psychiatric disorder including drug or alcohol dependence (as per SCID for DSM-5) except Nicotine Dependence
* Regular or current use of any prescription, herbal or illegal psychotropic medications in the past 1 year, with no current illegal drug use confirmed by urine toxicology (including cannabis)
* Drink more than 14 drinks per week for women or 21 drinks per week for men;
* Women who are pregnant or nursing
* Individuals who are currently taking medication that may affect cholinergic system or nicotine replacement therapy prescribed for smoking cessation;
* Contraindications to MRI such as claustrophobia or metal in their body, or to PET such as history of cancer Patient unlikely to be able to complete the study as determined by the PI or research assistants
* Blood donation within eight weeks of the start of the study
* History of a bleeding disorder or are currently taking anticoagulants (such as Coumadin, Heparin, Pradaxa, Xarelto)
* Known hypersensitivity to propylene glycol
* Planning to quit smoking with a set goal or time for quit attempt
* Untreated, unresolved acute pulmonary conditions (recurring bronchitis and Reactive airway disorder, as examples).
* Chronic symptoms on Health Questionnaire that would interfere with monitoring of vaping complication
* Naïve to vaping (vaping for less than 3 months and less than 12 times)

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12-30 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Brain beta-2 nicotinic acetylcholine receptor occupancy | 210 minutes
  PET Scan will be utilized to determine the brain beta-2 nicotinic acetylcholine receptor occupancy

SECONDARY OUTCOMES:
Maximum arterial blood nicotine | 90 minutes
  Arterial blood nicotine levels will be measured before, during, and after e-cig use.

CONTACTS AND LOCATIONS:
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-04-25): https://cdn.clinicaltrials.gov/large-docs/52/NCT04258852/ICF_000.pdf